CLINICAL TRIAL: NCT04862312
Title: VideoDining: Using Video Chat to Improve Nutritional Intake in Older Adults
Brief Title: Video Chat During Meals to Improve Nutritional Intake in Older Adults
Acronym: VideoDining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Foodnet Meals on Wheels (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011009963; 002254837 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2021-03-29; First posted 2021-04-27 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Malnutrition; Loneliness
Keywords: Older Adults; Geriatric; Elderly; Malnutrition; Nutrition; Video chat; Loneliness; Social Isolation; Social Facilitation of Eating; Aging in Place; Home Delivered Meals; Technology
MeSH Terms: conditions — Malnutrition; Social Isolation

STUDY DESIGN:
Intervention Model Description: All participants will receive the VideoDining intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VideoDine (Experimental): Use of video chat to eat a meal with a dining partner.
  Interventions: Behavioral: VideoDine

INTERVENTIONS:
Behavioral: VideoDine — Participants will VideoDine with a dining partner at least six times during an eight week period. VideoDining involves sharing a meal with someone not physically present using video chat technology. Dining partners will be recruited, trained and paired with participants. Participants will be provided Amazon Echo Show devices for video chat.

SUMMARY:
The VideoDining study is a Stage IB behavioral intervention development project. The objectives are to determine the feasibility and acceptability of using video chat during mealtimes (VideoDining) in community-dwelling older adults eating alone at home and to evaluate changes in nutritional intake and loneliness in response to VideoDining.

DETAILED DESCRIPTION:
The U.S. population is growing older and more adults are aging at home alone, by choice, or due to a lack of affordable senior housing. Older adults who live alone have a less healthy eating pattern, eat a smaller variety of foods and consume fewer fruits and vegetables than those living with others. Additionally, eating alone, social isolation and loneliness often accompany living alone and are independent risk factors for lower caloric intake, less variety in the diet and malnutrition. Community-based interventions are needed to improve the nutritional status of older adults living alone.

VideoDining uses video chat during mealtimes to virtually eat with another person and could provide social interactions and modeling to improve dietary intake in older adults eating alone. Extensive observational and experimental research shows that people eat more when dining with others than dining alone, called the social facilitation of eating. Additionally, a dining partner's modeling of eating can provide a guide for what and how much to eat. The investigators have conducted a Stage IA proof-of-concept study of VideoDining in older adults and will expand the development of this behavioral intervention with this study.

The goals are to determine the feasibility and acceptability of VideoDining and to evaluate changes in nutritional intake and loneliness in response to multiple VideoDining sessions in community-dwelling older adults eating alone at home. In this single-arm intervention study, thirty older adult Meals on Wheels participants will be scheduled to VideoDine with a dining partner six times. Using a mixed-methods approach, the investigators will collect data on older adults' ability to VideoDine, acceptance of VideoDining, dietary intake, and loneliness. Data will be collected before starting VideoDining, after each VideoDining session, and at the end of the study period. Development, adaptation and refinement of the VideoDining intervention are additional key outcomes of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Receive Meals-on-Wheels meals from Foodnet in Tompkins County, NY.
2. Aged 60-95 years old.
3. Consume Meals-on-Wheels meal alone.

Exclusion Criteria:

1. Non-English speaking.
2. Unable to read and write in English.
3. Inadequate vision and hearing to utilize video chat technology.
4. Unable cognitively to independently consent and participate in the study.
5. Already own and use an Amazon Echo Show.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change in caloric intake with VideoDining | 8 weeks
  A research interviewer will use video chat to collect three 24-hour dietary recalls with each participant prior to starting the VideoDining sessions (pre-VideoDining). During the intervention phase, a research interviewer will use video chat to collect a 24-hour dietary recall after each VideoDining session to capture dietary intake during the VideoDining meal and subsequent day (post-VideoDining). Change in dietary intake will be calculated by comparing average caloric intake on the three pre-VideoDining recalls to the average caloric intake on the final three post-VideoDining recalls.
Change in dietary intake pattern with VideoDining | 8 weeks
  A research interviewer will use video chat to collect three 24-hour dietary recalls with each participant prior to starting the VideoDining sessions (pre-VideoDining). During the intervention phase, a research interviewer will use video chat to collect a 24-hour dietary recall after each VideoDining session to capture dietary intake during the VideoDining meal and subsequent day (post-VideoDining). Change in diet quality will be determined by comparing average food group equivalents and the Healthy Eating Index (HEI) on the three pre-VideoDining recalls to the average for the final three post-VideoDining recalls.
Change in loneliness with VideoDining | 8 weeks
  The Revised 20-item UCLA Loneliness Scale and the 6-item De Jong Giervald Loneliness Scale will be collected prior to VideoDining and at the end of the study after VideoDining. The Revised 20-item UCLA Loneliness scale measures an individual's subjective feelings of loneliness and social isolation. Each question is scored 1-4, for a total of 20 to 80 points, with 80 indicating more loneliness. The 6-item De Jong Giervald Loneliness Scale uses a 3-item loneliness scale and a 3-item emotional scale. Each item is scored 0, 1 or 2, for a possible total score of 0-6, 0 being least lonely and 6 being most lonely. Total sum scores for each scale will be calculated pre and post VideoDining and compared.

SECONDARY OUTCOMES:
Feasibility: Enrollment rate | 12 months
  Number of people enrolled in the study as a percentage of people approached or who showed interest in the study during the recruitment time period.
Feasibility: Attrition | 12 months
  Percentage of enrolled participants who do not complete the study.
Feasibility: Completion rate | 8 weeks
  Percentage of participants who complete 6 or more VideoDining sessions in 8 weeks.
Feasibility: Technical assistance rate | 8 weeks
  Number of times participants require assistance to use video chat technology after initial training and set-up.
Acceptability: Acceptability of individual VideoDining sessions | 8 weeks
  Quantitative data from participant and dining-partner survey responses to questions on enjoyment, comfort, nervousness, technical issues, ease, and experience of VideoDining collected after each VideoDining session.
Acceptability: Acceptability of VideoDining | 8 weeks
  Qualitative data from end-of-study participant interviews and dining-partner focus groups. Participant responses to open ended questions about overall experience of VideoDining, use of videochat technology, and likes and dislikes of VideoDining will be coded and analyzed.
VideoDine Self-Efficacy | 8 weeks
  Participant responses to a single item survey question after each VideoDining session. Participant responses to survey questions about confidence level to perform the tasks of VideoDining, collected at the end of the study.
Social Support | 8 weeks
  Responses to the four questions on the Social Interaction Subscale of the Duke Social Support Index and one question about social interaction with friends and family using videochat will be collected prior to VideoDining and at the end of the study after VideoDining. The results will be compared pre and post VideoDining.

OTHER OUTCOMES:
Participant Hand Grip Strength | Baseline
  A nutrition professional will measure participant hand grip strength using the Jamar Hydraulic Hand Dynamometer at the participant's home. Measurements will be categorized using hand-grip strength cut-points for muscle weakness by gender and age (J Am Geriatr Soc. 2020 Jul;68(7):1429-1437.) and cut-points for likelihood of mobility limitation (J Am Geriatr Soc. 2010 Sep;58(9):1721-6).
Risk for Sarcopenia | Baseline
  A nutrition professional will administer the Strength, Assistance with Walking, Rising from a Chair, Climbing Stairs and Falls (SAR-F) survey. Outcomes of the SARC-F will be combined with calf circumference measured in question R (Calf Circumference in cm) of the MNA-FF to complete the SAR-CalF. A total sum score will be calculated, and participants categorized as at risk for sarcopenic (score 11-20) or non-sarcopenic (score 0-10). Results of the SAR-CalF will be combined with hand grip strength data and participant age and BMI to determine overall sarcopenia risk.
Risk of Malnutrition | Baseline
  A nutrition professional will administer the Mini Nutritional Assessment Full Form (MNA-FF). A total sum score will be calculated and categorized as Normal nutritional status (24-30 points), At risk of Malnutrition (17-23.5 points) and Malnourished (less than 17 points).
Participant Muscle Wasting | Baseline
  A trained nutrition professional will assess temporal, clavicular, calf and interosseous muscle wasting following the Academy of Nutrition and Dietetics Nutrition Focused Physical Exam guidelines. Muscle mass will be categorized at each site as: adequate (no wasting noted), mild, moderate or severe wasting.
Participant Subcutaneous Fat Wasting | Baseline
  A trained nutrition professional will assess orbital and triceps subcutaneous fat wasting following the Academy of Nutrition and Dietetics Nutrition Focused Physical Exam guidelines. Subcutaneous fat will be categorized at each site as: adequate (no wasting noted), mild, moderate or severe wasting.
Participant Weight | Baseline
  Participant weight will be measured using the Seca 869 Portable Scale. The participant will be weighed in their home while wearing light clothing and no shoes.
Participant Height | Baseline
  Participant height will be measured using the Seca 213 Portable Stadiometer at the participant's home.
Body Mass Index | Baseline
  Participant BMI will be calculated as weight in kilograms over height in meters squared using collected weight and height measurements.
Adequacy of Energy Intake | Baseline
  Participant energy needs will be calculated using the Mifflin St. Jeor formula using the collected height, weight and age data. Participant's average daily calorie intake will be determined from the three baseline 24-hour food recalls entered into ASA24. Adequacy of energy intake will be represented as a percentage of participant calculated intake out of calculated total estimated needs.
Weight Loss | Baseline
  Participant weight loss over the last 3 months will be assessed by the MNA-FF survey Question B (weight loss over the last 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Barre, MD, RDN, Principal Investigator — Cornell Univ
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the results will be shared within one year of final data collection and be available for at least 5 years. Data will be available on Open Science Framework. Access to the data will be granted upon request, after verification of the requesting investigator/clinician. Requests should be directed to LKB35@cornell.edu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available within one year of completion of data collection and be available for at least 5 years.
Access Criteria: Available upon request and verification of requesting investigator/clinician.